CLINICAL TRIAL: NCT05334238
Title: A Multi Center, Randomized, Controlled Clinical Study of the Efficacy and Safety of Orelabrutinib Maintenance Therapy After ASCT in Patients With Primary Central Nervous System Lymphoma
Brief Title: Orelabrutinib Maintenance Therapy After ASCT in Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCNSL-001
Record Dates: First submitted 2022-01-10; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Primary Central Nervous System Lymphoma; Orelabrutinib
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orelabrutinib (Experimental): oral administration of Orelabrutinib 150mg daily for 1 year, beginning 8 weeks after autologous transplantation
  Interventions: Drug: Orelabrutinib
- No Orelabrutinib (No Intervention): no treatment after autologous transplantation

INTERVENTIONS:
Drug: Orelabrutinib — oral administration of Orelabrutinib 150mg daily for 1 year, beginning 8 weeks after autologous transplantation
  Arms: Orelabrutinib

SUMMARY:
A multicenter, randomized, prospective clinical study of the efficacy and safety of Orelabrutinib maintenance therapy after Autologous Stem Cell Transplantation (ASCT) in patients with primary central nervous system lymphoma.

DETAILED DESCRIPTION:
This trial was designed as a multicenter, randomized controlled, prospective clinical study. To evaluate the efficacy and safety of Orelabrutinib maintenance therapy with ASCT in patients with primary lymphoma of the central nervous system in a prospective clinical study.

174 patients were enrolled in this study, and randomly divided into Orelabrutinib maintenance group experimental group or observation group (control group) by 1:1. The trial included a screening period (day -28 to day -1), a treatment period (oral administration of Orelabrutinib 150mg daily for 1 year, beginning 8 weeks after autologous transplantation), and a follow-up period (1 year after the end of the last treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18-65;
2. Primary CNS lymphoma patients with CR were evaluated in the final stage of first-line therapy, and the virus-infected patients were balanced between the experimental and control groups;
3. Laboratory tests (blood routine, liver and kidney function) meet the following requirements:

   A) Blood routine examination: white blood cell count ≥3.0×109/L, absolute neutrophil count ≥1.5×10^9/L, hemoglobin ≥90g/L, platelet ≥75×10^9/L; B) Liver function: transaminase ≤2.5× upper limit of normal value, bilirubin ≤1.5× upper limit of normal value; C) Renal function: serum creatinine 44-133 mmol/L;
4. Participants' ECOG physical status score was 0-2; The subject or his/her legal representative must provide written informed consent prior to conducting a special study examination or procedure.

Exclusion Criteria:

Presence of any of the following criteria will exclude a patient from enrollment:

* Uncontrolled cardio- and cerebro-vascular disease, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

  1. Neutrophils<1.5×10^9/L
  2. Platelets<80×10^9/L (Platelets<50×10^9/L in case of bone marrow involvement)
  3. ALT or AST is 2 times higher than the upper limits of normal (ULN), AKP and bilirubin are 1.5 times higher than the ULN.
  4. Creatinine is 1.5 times higher than the ULN or eGFR is lower than 40ml/min/1.73m^2 (according to Cockcroft-Gault Equation or MDRD Equation).
* HIV-infected patients
* Left ventricular ejection fraction<50%
* Patients with HbsAg positive are required to have HBV DNA<1.0×10^3 IU/ml before entering the group. In addition, if the patient is HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA test is also required, and HBV DNA<1.0×10^3 IU/ml is required before entering the group.
* Other anti-tumor treatments (lymphoma or other types of tumors) are currently in progress.
* Patients with psychiatric disorders or patients who are known or suspected to be unable to fully comply with the study protocol
* History of stroke or intracranial hemorrhage within 6 months prior to start of therapy
* Inability to swallow capsules or presence of diseases that significantly affect gastrointestinal function, such as malabsorption syndrome, post-bariatric surgery, inflammatory bowel disease and complete or incomplete intestinal obstruction
* Other medical conditions determined by the researchers that may affect the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival at 2 years | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Complete response rate at 1 years | Baseline up to data cut-off (up to approximately 1 years)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Overall survival at 2 years | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No